CLINICAL TRIAL: NCT06434571
Title: Comparing Telehealth-Delivered Cognitive Behavioral Therapy for Insomnia to Web-Based to Enhance Sleep, Reduce Fatigue, and Promote Neuroprotection
Brief Title: Comparing Telehealth-Delivered CBT-I to Web-Based CBT-I to Enhance Sleep, Reduce Fatigue, and Promote Neuroprotection
Acronym: CLEAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Catherine Siengsukon, PT, PhD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00160591
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis; Insomnia
Keywords: Cognitive behavioral therapy for insomnia; CBT-I
MeSH Terms: conditions — Multiple Sclerosis; Sleep Initiation and Maintenance Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telehealth cognitive behavioral therapy for insomnia (tCBT-I) (Experimental): 1x/week, 6-week 45-60 min one-one-one manualized program via video conferencing (HIPAA-compliant Zoom) with a trained research assistant that includes time in bed restriction, stimulus control, relaxation strategies, cognitive restructuring, and sleep health promotion education.
  Interventions: Behavioral: Telehealth cognitive behavioral therapy for insomnia (tCBT-I)
- Web-based cognitive behavioral therapy for insomnia (wCBT-I) (Experimental): The Go!ToSleep online program is a 6-week interactive, web-based program that delivers typical CBT-I treatment techniques of stimulus control, sleep restriction, behavioral modifications, relaxation techniques and cognitive restructuring with daily lessons (41 lessons in total)
  Interventions: Behavioral: Web-based cognitive behavioral therapy for insomnia (wCBT-I)
- Treatment as usual (TAU) (Other): The treatment as usual comparison group will be encouraged to continue with their usual care recommended by their physician and their usual activities and sleep habits during the period between baseline and 6-month reassessment.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Telehealth cognitive behavioral therapy for insomnia (tCBT-I) — The general sessions outlines are as follows with each session:
  Session 1: determine treatment plan, set up sleep schedule and stimulus control, discuss strategies for how to stay awake to prescribed hour and what to do if wake up in middle of night, sleep hygiene education Session 2: continue upward titration of total sleep time, review sleep hygiene; introduce diaphragmatic breathing Session 3: continue upward titration of total sleep time, introduce mindfulness Session 4: continue upward titration of total sleep time, introduce progressive muscle relaxation Session 5: continue upward titration of total sleep time, discuss negative sleep beliefs Session 6: assess global treatment gains, discuss relapse prevention
  Arms: Telehealth cognitive behavioral therapy for insomnia (tCBT-I)
Behavioral: Web-based cognitive behavioral therapy for insomnia (wCBT-I) — Participants receive a daily e-mail reminder to access the program and to complete a sleep log for the prior night's sleep. After completing the sleep log, the daily lesson is made available. Each participant will be provided with a unique password to access the online program.
  Arms: Web-based cognitive behavioral therapy for insomnia (wCBT-I)
Behavioral: Treatment as usual (TAU) — They will be encouraged to avoid starting any new treatment for their sleep unless recommended by their physician. They will be offered access to the web-based CBT-I program following the 6-month reassessment to complete if they wish.
  Arms: Treatment as usual (TAU)

SUMMARY:
The objective of this RCT is to assess the efficacy of one-on-one telehealth CBT-I (tCBT-I) compared to web-based CBT-I (wCBT-I) and treatment as usual (TAU) to improve sleep outcomes (Aim 1), fatigue and quality of life (Aim 2), and promote neuroprotection (Exploratory Aim 3), and to explore the characteristics of participants that predict improvement in sleep outcomes (Exploratory Aim 4). Reassessment of outcomes will be completed after the 6-week intervention and 6 months following completion of interventions.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Diagnosis of relapsing-remitting or secondary progressive MS based on established guidelines21 and verified by their neurologist
* Mild-to-moderately severe disability (≤ 6 on Patient Determined Disability Steps (PDDS) scale)
* Report of difficulty falling asleep, maintaining sleep, or waking up too early at least 3 nights/week for the past 3 months with significant distress and impact on function despite adequate opportunity for sleep and not due to other sleep disorders as indicated in the DSM-5
* ≥10 on Insomnia Severity Index
* English speaking
* ≥31 on Telephone Interview of Cognitive Status
* Has a high school diploma or equivalent to serve as a proxy measurement of reading ability to ensure adequate reading ability to participate in the study
* Report having access to internet service or a data plan and access to a computer, tablet, or smart phone

Exclusion Criteria:

* Known untreated sleep disorder (such as sleep apnea or restless legs syndrome)
* >3 on STOP BANG indicating increased risk of sleep apnea
* Restless legs syndrome as determined by RLS-Diagnosis Index
* Circadian rhythm sleep-wake disorder as determined by the Sleep Disorders-Revised
* Parasomnia as determined by the Sleep Disorders-Revised
* If taking benzodiazepines, non-benzodiazepines, or melatonin supplements or agonists for insomnia, taking < 3 months or dose has changed in past 3 months
* Score of ≥20 on the Patient Health Questionnaire (PHQ-9) indicating severe depression or endorsement of suicidal ideation (answer 1, 2 or 3 on #9 of the PHQ-9)
* Score of ≥15 on the Generalized Anxiety Disorder (GAD-7) indicating severe anxiety
* Current or history (up to 2 years) of alcohol or drug or alcohol abuse as indicated by DSM-5 criteria
* History of other nervous system disorder such as stroke or Parkinson's disease
* Currently pregnant or intending to become pregnant in the next 6 months
* Severe mental illness such as schizophrenia or bipolar disorder
* Severe neurological or sensory impairments that would interfere significantly with testing
* Relapse and/or corticosteroid use in the past 8 weeks
* History of (within 5 years) or currently conducting overnight shift work including hours of midnight-4am
* Currently receiving a behavioral sleep health intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | baseline, Week 6, Week 12
  The ISI consists of 7 questions, each rated on a 0-4 scale. The range of scores on the ISI is 0-28, with a score of ≥ 10 suggesting clinical insomnia. The lower the score the less severe insomnia.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | baseline, Week 6, Month 6
  The PSQI consists of 9 items within 7 sleep categories. The 7 sleep category scores are summed to form a single global score ranging from 0-21. A global score of >5 reflects poor sleep quality.
Epworth Sleepiness Scale (ESS) | baseline, Week 6, Month 6
  Consists of eight scenarios of daily activity, and participants use a four-point Likert scale to rate how likely they are to doze. Score ranges 0-24 with a higher score indicating daytime sleepiness.
Dysfunctional Beliefs About Sleep | baseline, Week 6, Month 6
  This assessment is a 10 item Likert-scale self-report questionnaire. Higher scores indicate more dysfunctional beliefs.
Positive Affect and Negative Affect Schedule (PANAS) | baseline, Week 6, Month 6
  The PANAS is a 20-item self-report questionnaire used to measure positive and negative emotions. There are two subscales (Positive Affect and Negative Affect) with 10 items each. The respondent scores how applicable a list of emotions are on a 5-point Likert scale with 1 = "Very slightly or not at all" to 5 = "Extremely". A higher score on the Positive Affect subscale indicates greater intensity of positive emotions, and a high score on Negative Affect indicate greater intensity of negative emotions.
Sleep Self-Efficacy Scale (SESS) | baseline, Week 6, Month 6
  The SESS is a 9 item self-report Likert-scale questionnaire use to identify sleep self-efficacy. Scores range from 0-45 and a higher score indicates higher sleep self-efficacy.
Actigraphy | baseline, Week 6, Month 6
  Participants will wear an actigraph on their non-dominant wrist for 7 nights to assess sleep/wake cycle. Mains variables of interest are sleep regularity, timing, efficiency, and duration
Modified Fatigue Impact Scale (MFIS) | baseline, Week 6, Month 6
  The MFIS assesses the impact of fatigue on daily activities for the month prior. The MFIS consists of 21 items with 3 subscales: physical, cognitive, and psychosocial. The score on the 21 items are scored with a range of 0-84 with a higher score indicating a greater impact of fatigue.
Fatigue Severity Scale (FSS) | 'baseline, Week 6, Month 6
  The FSS assesses the impact of fatigue on activities for the week prior and consists of 9 questions. The mean of the 9 scores is calculated with a range of 0-7.
Multiple Sclerosis Impact Scale (MSIS-29) | baseline, Week 6, Month 6
  Quality of life will be assessed using the Multiple Sclerosis Impact Scale (MSIS-29). MSIS-29 is total of 29 items scale, with subscales of physical (20 items) and psychological (9 items). Responses computed in a range from 0-100, and higher scores indicating a worse quality of life due to physical and physiological impacts of MS
Cognitive Failures Questionnaire (CFQ) | baseline, Week 6, Month 6
  The CFQ assesses perception of cognitive abilities over the past 6 months. consists of 25 items that the individual rates on a 5-point Likert scale with 0 = "never" and 4 = "Very Often" with a summary score of 0-100 with a higher score indicating poorer perceived cognitive abilities.
plasma neurofilament light (NfL) | baseline, Week 6, Month 6
  blood marker of axonal damage

OTHER OUTCOMES:
Patient-Determined Disability Steps (PDDS) | baseline
  Disability will be assessed using the PDDS scale which is a single-item 9 point scale ranging from "normal" (score of 0) to "bedridden" (score of 8).
Patient Health Questionnaire (PHQ-9) | baseline, Week 6, Month 6
  Depressive symptoms will be assessed using the 9-item Patient Health Questionnaire (PHQ-9), with a score of ≥20 suggesting severe depression. It consists of 9 items with a score ranging from 0-27.
Generalized Anxiety Disorder Assessment (GAD-7) | baseline, Week 6, Month 6
  Anxiety symptoms will be assessed using the 7-item GAD-7, with a score of ≥15 indicating severe anxiety. This questionnaire consists of 7 items, and the score from each item is summed for an overall score ranging from 0-21 with a higher score indicating a higher level of anxiety
Adherence to CBT-I intervention | Each CBT-I session Week 1-6
  To assess adherence to the CBT-I intervention, the sleep log will be used to assess number of mornings/week got out of bed at agreed upon time and the number of times got out of bed if unable to sleep. A total percentage will be calculated and used as the outcome of interest.
Diet quality | baseline
  Participants will be asked "In general, how healthy is your overall diet?" and will rate on a 5-point Likert scale (5 = "excellent", 4 = "very good", 3 = "good", 2 = "fair", 1 = "poor")
Eating regularity | baseline, Week 6, Month 6
  Participants will mark on the sleep log at each assessment period the time period for eating breakfast, lunch, and dinner. Variability in mealtime will be quantified as the standard deviation from the individual's mean meal start time.
Nighttime urination frequency | baseline, Week 6, Month 6
  Participants will mark on the sleep log the number of times they wake up to void their bladder during the sleep opportunity window.
PainDetect | baseline, Week 6, Month 6
  PainDetect includes 13 items that assesses neuropathic pain. A total score ranges from -1 to 38, with higher scores indicating higher levels of neuropathic pain.
Fibromyalgia Survey Questionnaire | baseline, Week 6, Month 6
  Fibromyalgia Survey Questionnaire includes the assessment of the number of painful body regions. Scores ranges from 0-31. A higher score indicates worse symptoms.
PROMIS SF v.1.0 - Pain Intensity | baseline, Week 6, Month 6
  Measures max and average pain intensity during past 7 days. The T-score value, with a mean of 50 and standard deviation of 10 representing the rescaled raw score, will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center- Sleep, Health and Wellness Laboratory, Kansas City, Kansas, United States